CLINICAL TRIAL: NCT06814184
Title: Improving Glycemic Control Among Underserved Patients With Insulin-treated Type 2 Diabetes Through Nurse-led, App-based Behavioral Intervention
Brief Title: Virtual Diabetes Care for Low Socioeconomic Status Adults With Type 2 Diabetes on Insulin Therapy
Acronym: virtual care
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Helen NC Chen PhD, FNP, PHD RN CRNP, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: Pro2025000096; K99NR020377 (NIH)
Record Dates: First submitted 2025-02-01; First posted 2025-02-07 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Type 2 Diabetes
Keywords: diabetes app; behavioral intervention; self-management; diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: Clinic 1 starts enrollment and intervention on 1/2/2026, while Clinic 2 starts enrollment but intervention starts on 4/1/2026. We cannot deliver intervention the same time rallel step-wedge, give two clinics intervention can't deliver intervention same time
Who Masked: Participant
Masking Description: Both clinics collect baseline at the same time for both clinics. Masking participants that we tell participants that we will reach out to when intervention rolls out. Clinic 2 will roll out 3 months later than Clinic 1.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental with intervention (Experimental): Intervention starts at enrollment
  Interventions: Behavioral: app-based nurse-led virtual diabetes care
- Delayed Intervention (Other): Intervention delivery 3 months after enrollment
  Interventions: Behavioral: app-based nurse-led virtual diabetes care

INTERVENTIONS:
Behavioral: app-based nurse-led virtual diabetes care — A nurse-led, app-based behavioral intervention consisting of (1) education via MyChart messaging, (2) problem solving with an action plan via phone, and (3) remote patient monitoring via mySugr app to identify the need to adjust treatment

SUMMARY:
This 12-month pilot tests a nurse-led, app-based intervention to improve diabetes self-management for low-socioeconomic status patients. It includes MyChart messing to give education, phone help on problem-solving with clinicians, and using a diabetes app to track data. The study aims to enhance self-management behaviors through health technology.

DETAILED DESCRIPTION:
Guided by the Self- and Family Management Framework, which specifies facilitators and barriers to self- management behaviors, this project tests strategies for delivering virtual diabetes care to help low-socioeconomic status patients and clinicians use health information technology to support self-management behaviors. It is a 12-month pilot nurse-led, app-based behavioral intervention consisting of three evidence-based interventions: (1) education on A1C results and goal-setting via MyChart, the Epic electronic health record's patient portal; (2) a problem-solving action plan developed collaboratively by clinicians and patients; and (3) remote monitoring via mySugr, a top- rated diabetes app, to track blood glucose and identify the need for treatment adjustments.

ELIGIBILITY:
Inclusion Criteria:

* A1C>8% within 12 months prior baseline
* A1C>8% at baseline
* Low-SES (defined as a Medicaid recipient or dual Medicaid and Medicare recipient or self-reported low income based on National Poverty Guidelines)
* Age 18 or older
* Type 2 diabetes
* On insulin therapy
* Owning and using Android or iOS smartphone for at least 6 months
* English proficiency
* Adequate vision to read text messages on their current smartphone
* Smartphone use proficiency. Smartphone proficiency will be self-reported and determined by telephone as the ability to use a smartphone in ways other than emailing, texting, and making phone calls.

Exclusion Criteria:

* Pregnancy
* Patients with cognitive impairment who will be screened with the Six-Item Screener to Identify Cognitive Impairment Among Potential Research Subjects.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-01-02 (Estimated); Primary Completion 2028-01-03 (Estimated); Study Completion 2028-04-03 (Estimated)

PRIMARY OUTCOMES:
Glycemic control: glycated hemoglobin AIC | baseline, 3, 6, 9, and 12 months
  Electronic health record extracted lab test drawn at baseline, 3, 6, 9, and 12 months
Glycemic control - the rate of pre-prandial blood glucose readings in target range | baseline, 3, 6, 9, and 12 months
  Home monitoring glucometer at baseline and diabetes app report containing blood glucose readings at home for 3, 6, 9, and 12 months. It is calculated from the number of BG that met the target divided by the total number of BG tested.
Glycemic control - the rate of peak postprandial blood glucose reading in target range | baseline, 3, 6, 9, and 12 months
  Blood glucose reading obtained from patient's home monitoring glucometer at baseline and diabetes app report containing blood glucose readings at home for 3, 6, 9, and 12 months. It is calculated from the number of BG that met the target divided by the total number of BG tested.

SECONDARY OUTCOMES:
Diabetes Knowledge Test 2 (23 iems) for knowledge change | baseline, 3, 6, 9, and 12 months
  This scale assesses the knowledge of individuals regarding diabetes management and self-care. 0 is minimal and 23 is maximal. Higher is better outcome reflecting high knowledge.
Diabetes Empowerment Scale Short 28 items for self-efficacy change | baseline, 3, 6, 9, and 12 months
  The DES-28 has been validated and is considered a reliable tool for assessing the psychosocial aspects of diabetes management, making it useful for various educational and psychosocial interventions related to diabetes. 28 is minimal, 140 is max. Higher is better outcome, reflecting greater empowerment and self-efficacy in managing diabetes.
AHC Health-Related Social Needs Screening Tool (10 items) for Social Determinants of Health Change | baseline, 3, 6, 9, and 12 months
  It help healthcare providers identifies the social needs of their patients, which can inform interventions and resource allocation. 0 is minimal, 10 is max. Higher score is greater number of identified health-related social needs, which may suggest worse outcomes in terms of social determinants of health.
Jalowiec Coping Scale 40 items for coping style and effectiveness change | baseline, 3, 6, 9, and 12 months
  The scale evaluates both problem-oriented and affective-oriented coping strategies, providing insights into how individuals manage the challenges associated with diabetes. 40 is minimal, 200 is max. Higher score indicate a greater use of coping strategies, which generally suggests better coping and potentially better outcomes in managing diabetes.
Diabetes Distress Scale (17 items) for quality of life change | baseline, 3, 6, 9, and 12 months
  It measures the emotional stress specific to diabetes management. a valuable tool for identifying patients who may need additional support in managing the emotional burdens associated with diabetes. 17 is minimal, 102 is max. Higher score indicates greater levels of diabetes distress, which generally suggests worse outcomes in terms of emotional well-being and diabetes management.
Summary of Diabetes Self-Care Activities Measure (11 items) for Self-management activity changes | baseline, 3, 6, 9, and 12 months
  It is a reliable and valid tool for evaluating diabetes self-management behaviors and is useful in both research and clinical settings. 0 is minimal indicating no self-care activities performed, 11 is max indicating all self-care activities performed. Higher score indicate Measure consists of 11 items that assess various aspects of diabetes self-management.
BG testing frequency change | baseline, 3, 6, 9, and 12 months
  The number of blood glucose readings obtained from patient's home monitoring glucometer at baseline and the number of blood glucose readings listed in the diabetes app report at home for 3, 6, 9, and 12 months.
Diabetes Numeracy Test short (15 items) for knowledge change | baseline, 3, 6, 9, and 12 months
  This test assesses diabetes-related numeracy skills that are essential for effective self-management of diabetes, such as interpreting blood glucose readings and calculating carbohydrate intake. 0-15, 0 is minimal with no correct answer, 15 is max. Higher is better outcome reflecting higher numeracy.

CONTACTS AND LOCATIONS:
Overall Officials: Helen NC Chen, PhD, Principal Investigator — Rutgers School of Nursing

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared. Each participant will be given a unique study identification number that will be used on all study forms and data files. Each participant's identifying data will be separated from the study data. All data will be de-identified with a participant code number. The code linking a participant to their code number will be maintained in a separate file on a secure server at Rutgers (e.g., Microsoft Teams, Box).